CLINICAL TRIAL: NCT03266471
Title: Cytokines and Genes in Therapeutic Response in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Scoville, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 171198
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Cytokines; Pharmacogenetics
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any remaining serum or tissue samples may be evaluated for other markers of IBD or stored for future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease Patients: Patients that are seen in the Inflammatory Bowel Disease clinic with CD confirmed by endoscopy or radiology assessment who are initiating either an anti-tumor necrosis factor (TNF)-α agent (infliximab, adalimumab, certolizumab, or infliximab biosimilar), ustekinumab, or vedolizumab as part of their routine clinical care will be asked to provide blood samples, stool samples, and intestinal biopsies from standard of care colonoscopy at baseline and post therapy of at least 6 weeks duration but not more than 52 weeks.
  Interventions: Diagnostic Test: Baseline blood sample; Diagnostic Test: Baseline intestinal biopsies; Other: Crohn's disease activity index (CDAI); Diagnostic Test: Post treatment blood sample; Diagnostic Test: Post treatment intestinal biopsies; Diagnostic Test: Baseline stool sample; Diagnostic Test: Post treatment stool sample
- Controls: Healthy adults without IBD undergoing colonoscopy for colorectal cancer screening or other non-IBD related indication will be asked to provide blood samples, stool samples and intestinal biopsies from standard of care colonoscopy.
  Interventions: Diagnostic Test: Baseline blood sample; Diagnostic Test: Baseline intestinal biopsies; Diagnostic Test: Baseline stool sample

INTERVENTIONS:
Diagnostic Test: Baseline blood sample — Blood sample for cytokine measurements and genetics.
Diagnostic Test: Baseline intestinal biopsies — Up to 20 additional biopsies will be obtained at the time of standard of care colonoscopy. It is not felt that additional biopsies substantially increases the risk of a colonoscopy. Cytokine measurements will be performed on the tissue collected.
Other: Crohn's disease activity index (CDAI) — To determine response, a Crohn's Disease Activity Index (CDAI) score will be obtained at time point 1 and time point 2 in all enrolled CD patients. The CDAI is a well validated symptom index for CD which assesses 8 factors including stool frequency, abdominal pain, general well being, CD complications, HCT, and deviation from ideal body weight.
  Groups: Crohn's disease Patients
Diagnostic Test: Post treatment blood sample — Blood sample for cytokine measurements after patients have been on therapy for at least 6 weeks but no more than 52 weeks.
  Groups: Crohn's disease Patients
Diagnostic Test: Post treatment intestinal biopsies — Up to 20 additional biopsies will be obtained at the time of standard of care colonoscopy at least 6 weeks but no more than 52 weeks after initiation of therapy. It is not felt that additional biopsies substantially increases the risk of a colonoscopy. Cytokine measurements will be performed on the tissue collected.
  Groups: Crohn's disease Patients
Diagnostic Test: Baseline stool sample — Stool sample for inflammatory markers or microbiome analysis.
Diagnostic Test: Post treatment stool sample — Stool sample for inflammatory markers or microbiome analysis.
  Groups: Crohn's disease Patients

SUMMARY:
Inflammatory bowel disease (IBD), consisting of two major forms, Crohn's disease (CD) and ulcerative colitis (UC), affects more than 1.6 million people in the United States alone. Though the precise mechanisms underlying the inflammation and immune responses in IBD are still being investigated, various inflammatory mediators, including pro-inflammatory cytokines, and genes have been implicated in the disease process. At present, there are no reliable mechanisms to predict response to individual IBD medications. The investigators seek to evaluate whether inflammatory cytokines change longitudinally during treatment with anti-cytokine agents in both treatment primary responders and primary non-responders. In addition, the investigators will be evaluating the pharmacogenetics of treatment response to these agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are seen in the Inflammatory Bowel Disease clinic with Crohn's disease who are initiating either treatment as part of their routine clinical care.
* Healthy adults without IBD undergoing colonoscopy for colorectal cancer screening or other non-IBD related indication.

Exclusion Criteria:

* pregnant
* have a known coagulopathy or bleeding disorder
* have known renal or hepatic impairment
* have a history of organ transplantation
* CD patients who are being seen in consultation and do not plan to receive longitudinal care through initiation their new therapy at the Vanderbilt IBD center will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for a colonoscopy at the Vanderbilt Endoscopy Laboratory as part of their routine care and who do not meet any of the pre-defined exclusion criteria will be considered for participation in the study as control subjects. Patients who are part of the Vanderbilt IBD practice who initiate therapy on an anti-TNF, ustekinumab, or vedolizumab as part of their routine care will be considered for participation in the study as subjects.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Compare longitudinal cytokine measurements in treatment responders versus nonresponders. | 52 weeks
  The investigators will classify Crohn's disease subjects as primary responders or primary non-responders to anti-TNF-α, ustekinumab, or vedolizumab therapy based on clinical, endoscopic, and/or histologic data. The investigators will compare serum and tissue cytokines in CD subjects at before and after treatment initiation.

SECONDARY OUTCOMES:
Compare serum and tissue pro-inflammatory cytokines in CD patients and healthy subjects. | 26 weeks
  The investigators will compare serum and tissue cytokine/chemokine levels to see if Crohn's disease patients express a difference versus control.
To assess whether gene variants are associated with treatment response. | 52 weeks
  The investigators will collect a one time whole blood sample from subjects starting a new anti-cytokine agent (infliximab, infliximab biosimilar, adalimumab, certolizumab, ustekinumab, or vedolizumab) and extract DNA and genotype. The investigators will look for associations between genotype and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Scoville, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Inflammatory Bowel Disease Clinic, Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No